CLINICAL TRIAL: NCT02816021
Title: Phase II Study of Oral Azacitidine (CC-486) in Combination With Pembrolizumab (MK-3475) in Patients With Metastatic Melanoma
Brief Title: Study of Oral Azacitidine (CC-486) in Combination With Pembrolizumab (MK-3475) in Patients With Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0069; NCI-2016-01185 (Other: NCI CTRP)
Record Dates: First submitted 2016-06-15; First posted 2016-06-28 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Melanoma and Other Malignant Neoplasms of Skin; Metastatic Melanoma
Keywords: Melanoma and other malignant neoplasms of skin; Metastatic melanoma; Advanced melanoma; Azacitidine; 5-azacytidine; 5-aza; Vidaza; 5-AZC; Ladakamycin; NSC-102816; Azacytidine; Pembrolizumab; Keytruda; MK-3475; SCH-900475
MeSH Terms: conditions — Melanoma | interventions — Azacitidine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Metastatic Melanoma - PD-1 Naive (Experimental): Thirty-six participants with metastatic melanoma that are PD-1 naïve enrolled in treatment Arm A.
  Treatment consists of 3-week cycles and continues until disease progression. Oral Azacitidine administered by mouth daily for 15 days (Days 1-15) of every cycle. Pembrolizumab administered by vein every 3 weeks and after the oral dose of Azacitidine on concurrent treatment days.
  Interventions: Drug: Azacitidine; Drug: Pembrolizumab
- Arm B: Metastatic Melanoma - Post PD-1 Progression (Experimental): Thirty-five participants with metastatic melanoma that have progressed on PD-1 directed therapy enrolled in treatment Arm B.
  Treatment consists of 3-week cycles and continues until disease progression. Oral Azacitidine administered by mouth daily for 15 days (Days 1-15) of every cycle. Pembrolizumab administered by vein every 3 weeks and after the oral dose of Azacitidine on concurrent treatment days.
  Interventions: Drug: Azacitidine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Azacitidine — 300 mg by mouth daily for 15 days (Days 1-15) of every cycle.
  Other Names: 5-azacytidine; 5-aza; Vidaza; 5-AZC; Ladakamycin; NSC-102816; Azacytidine
Drug: Pembrolizumab — 200 mg by vein every 3 weeks and after the oral dose of Azacitidine on concurrent treatment days.
  Other Names: Keytruda; MK-3475; SCH-900475

SUMMARY:
You are being asked to take part in this study because you have advanced melanoma.

The goal of this clinical research study is to learn if oral azacitidine (CC-486) and pembrolizumab (MK-3475) can help to control melanoma. The safety of this drug combination will also be studied.

This is an investigational study. Azacitidine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS) and acute myeloid leukemia. Pembrolizumab is FDA approved and commercially available for the treatment of melanoma. It is considered investigational to use this drug combination to treat melanoma.

The study doctor will explain how the study drugs are designed to work.

Up to 71 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 3 weeks.

You will take azacitidine by mouth 1 time each day on Days 1-14 of each cycle. You may be asked to complete a Pill Diary for this drug. On this Pill Diary you will record the date, time, and number of azacitidine tablets you took that day. You will bring the Pill Diary to each Study Visit while you are on this drug.

You will receive pembrolizumab by vein over about 30 minutes on Day 1 of each cycle.

Study Visits:

On Day 1 of Cycles 1-3:

* You will have a physical exam.
* Blood (about 2½ teaspoons) will be drawn for routine tests.
* During Cycle 1 (if it was not done at screening) and Cycle 3, blood (about 1 teaspoon) will be drawn to learn if the study drugs have affected the disease.
* During Cycle 3 only, you will have 4 core needle tumor biopsies.
* If you can become pregnant, part of the above routine blood sample or urine will be collected for a pregnancy test.

On Day 1 of Cycle 4:

* You will have a physical exam.
* Blood (about 2½ teaspoons) will be drawn for routine tests and to learn if the study drugs have affected the disease.
* If you can become pregnant, part of the above routine blood sample or urine will be collected for a pregnancy test.

You will have an MRI or CT scan at the end of Cycle 4.

On Day 1 of Cycle 5:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and to check the status of the disease.
* You will have 4 core needle tumor biopsies.
* If you can become pregnant, part of the above routine blood sample or urine will be collected for a pregnancy test.

On Day 1 of Cycles 6 and beyond:

* You will have a physical exam.
* Blood (up to 3½ teaspoons) will be drawn for routine tests.
* If you can become pregnant, part of the above routine blood sample or urine will be collected for a pregnancy test.

At the end of Cycle 8 and then every 4 cycles after that (Cycles 12, 16, 20, and so on), you will have an MRI or CT scan.

Length of Study:

You may continue taking the study drugs for up to 24 months or 35 doses, whichever is later. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

End-of-Treatment Visit:

* Blood (about 4 teaspoons) will be drawn for routine testing and to learn how the study drug has affected the disease.
* You will have an MRI or CT scan.
* If you stop treatment because the disease got worse, you may have 4 core needle tumor biopsies.
* If you can become pregnant, part of the above routine blood sample or urine will be collected for a pregnancy test.

Follow-Up:

If you stopped taking the study drug for any reason other than the disease getting worse, you will have an MRI or CT scan every 12 weeks.

If the disease appears to get worse during this time, you may be eligible to be re-treated with pembrolizumab for an additional year (described below).

Re-Treatment:

If the disease got worse during follow-up and you are still eligible, you may be able to receive up to 1 year of additional treatment with pembrolizumab. If you continue to receive pembrolizumab, you will receive it at the same dose and schedule as described above. You will also continue to have study visits as described above.

Safety Follow-Up Visit:

About 30 days after your last dose of study drugs or before you start a new anti-cancer treatment (whichever happens first), you will have a safety follow-up visit. At this visit, you will have a physical exam and blood (about 2½ teaspoons) will be drawn for routine tests.

This may mean that you have 2 safety follow-up visits if you receive an additional year of pembrolizumab.

Long-Term Follow-Up:

After follow-up, you will be called every 12 weeks by a member of the study staff to learn how you are doing. This call should last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have unresectable Stage III through stage IV metastatic melanoma that have not received prior PD-1 directed therapy (Arm A) or that have progressed despite prior PD-1 directed therapy (Arm B).
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be >/= 18 years of age on day of signing informed consent.
4. Have measurable or evaluable disease based on RECIST 1.1.
5. Be willing to provide archival or fresh tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1. Subjects from whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Principal Investigator.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation. Hematological: Absolute neutrophil count (ANC) >/= 1,500 /mcL; Platelets >/= 100,000 / mcL; Hemoglobin >/= 9 g/dL or >/= 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment). Renal: Serum creatinine </= 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >/= 60mL/min for subjects with creatinine levels > 1.5 X ULN. Hepatic: Serum total bilirubin </= 1.5 X ULN or direct bilirubin </= ULN for subjects with total bilirubin levels > 1.5 ULN; AST (SGOT) and ALT (SGPT) 9 </= 2.5 X ULN OR </= 5 X ULN for subjects with liver metastases.
8. contd from #7. Albumin >/= 2.5 g/dL. Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) </=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants </= 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab, azacitidine, mannitol, or any of their excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Significant active cardiac disease within the previous 6 months including: - NYHA class 4 CHF - Unstable angina - Myocardial infarction
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent [for Arm A only].
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate in Participants with Metastatic Melanoma That Are PD-1 Naïve (Arm A) or That Have Progressed on PD-1 Directed Therapy (Arm B) | After 4 cycles. Each cycle is 21 days.
  Objective Response Rate determined by Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
Objective Response Rate in Participants with Metastatic Melanoma That Are PD-1 Naïve (Arm A) or That Have Progressed on PD-1 Directed Therapy (Arm B) | After 4 cycles. Each cycle is 21 days.
  Objective response rate determined by Immune Related Response Criteria (ir-RC).

SECONDARY OUTCOMES:
Overall Survival in Participants with Metastatic Melanoma That Are PD-1 Naïve (Arm A) or That Have Progressed on PD-1 Directed Therapy (Arm B) | 1 year
  Overall survival defined as the interval between time of enrollment and the date of death from any cause. Overall survival analyzed using the Kaplan-Meier method.
Progression Free Survival in Participants with Metastatic Melanoma That Are PD-1 Naïve (Arm A) or That Have Progressed on PD-1 Directed Therapy (Arm B) | After 6 cycles. Each cycle is 21 days.
  Progression free survival defined as the time between the date of enrollment and the date of either disease progression or date of death, whichever is earlier. Progression free survival summarized and plotted using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Tawbi, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org